CLINICAL TRIAL: NCT02657577
Title: REseArCH INteGration in Women, Infants, and Children: REACHING WIC
Brief Title: REseArCH INteGration in Women, Infants, and Children
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Leanne Redman, Principal Investigator, Pennington Biomedical Research Center
Other Study IDs: PBRC 2014-048
Record Dates: First submitted 2016-01-14; First posted 2016-01-18 (Estimated); Results first posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2022-09

CONDITIONS: Body Weight Changes
Keywords: Women; Infants and Children; Survey
MeSH Terms: conditions — Body Weight Changes

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- WIC staff: WIC staff is eligible to complete the WIC staff online survey if the individual is at least 18 years of age and have been employed at a WIC Clinic or DHH in Louisiana for at least 6 months in the past 2 years.
  Interventions: Other: There is no intervention
- WIC clients: WIC client is eligible to complete the WIC client online survey if the individual is at least 18 years of age and received WIC services during pregnancy or postpartum or have had a child who received WIC services in the past 2 years.
  Interventions: Other: There is no intervention

INTERVENTIONS:
Other: There is no intervention — There is no intervention

SUMMARY:
WIC is a governmental program that provides healthy foods, nutrition education and referrals to other health and social services. With the goal of applying for a future grant to expand the dissemination of SmartLoss® within the WIC program, feedback from WIC staff and WIC clients must be solicited to better understand the burden and barriers of integrating these kinds of programs and with WIC participants.

DETAILED DESCRIPTION:
Participants will complete a 15 minute online survey. WIC Staff will be eligible to complete the WIC staff survey and WIC clients will be eligible to complete the WIC client survey. This is a qualitative research study designed to identify the receptiveness of implementing a weight management program in the WIC program and the barriers to weight management intervention as described by WIC staff and WIC clients.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are at least 18 years old
* Have been employed or volunteered at a WIC Clinic or DHH in Louisiana for at least 6 months in the past 2 years OR received WIC services during pregnancy or postpartum or have had a child who received WIC services in the past 2 years

Exclusion Criteria:

* Less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 1000 individuals will be identified at WIC clinics in Louisiana. Participants must be at least 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 628 (Actual)
Dates: Start 2016-02-03 (Actual); Primary Completion 2016-06-02 (Actual); Study Completion 2016-06-02 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | WIC Staff | WIC Clients
Started | 201 | 427
Completed | 164 | 383
Not Completed | 37 | 44

BASELINE CHARACTERISTICS:
Population: In the WIC clients survey, age, sex, and race were collected categorically. The WIC staff survey did not ask any identifying or demographic questions so age, sex, and race were not collected in the WIC staff surveys.
Groups:
- Total: Total of all reporting groups
Arm/Group | WIC Staff | WIC Clients | Total
Number analyzed (Participants) | 164 | 383 | 547
Age, Customized [Count of Participants; unit: Participants]
  Age (Categorical): Between 18 and 29 years | 0 | 203 | 203
  Age (Categorical): Between 30 and 39 years | 0 | 76 | 76
  Age (Categorical): Older than 39 years | 0 | 17 | 17
  Age (Categorical): Unanswered | 0 | 87 | 87
  Age (Categorical): Not Collected | 164 | 0 | 164
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex/Gender: Female | 0 | 383 | 383
  Sex/Gender: Male | 0 | 0 | 0
  Sex/Gender: Not Collected | 164 | 0 | 164
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 0 | 140 | 140
  Race: Black or African American | 0 | 179 | 179
  Race: Asian | 0 | 5 | 5
  Race: American Indian | 0 | 10 | 10
  Race: Native Hawaiian or Pacific Islander | 0 | 2 | 2
  Race: Other | 0 | 46 | 46
  Race: Unanswered | 0 | 1 | 1
  Race: Not Collected | 164 | 0 | 164

OUTCOME MEASURES:

1. Primary Outcome: Receptiveness to Weight Management Interventions in the WIC Program
Description: WIC staff and WIC clients were asked if they were receptive to implementing weight management interventions in the WIC program with answer options: Yes, No, Neutral, or Unanswered.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | WIC Staff | WIC Clients
Number analyzed (Participants) | 164 | 383
Participants
  Yes | 126 | 184
  No | 6 | 190
  Neutral | 30 | 0
  Unanswered | 2 | 9

2. Primary Outcome: Barriers to WIC Appointments as Described by WIC Clients
Description: WIC clients were asked what are barriers that they experience attending their WIC appointments.
Time Frame: 1 day
Population: This question was only asked as part of the WIC clients survey as it dealt directly with barriers that WIC Clients experience.
Measure: Count of Participants; unit: Participants
Arm/Group | WIC Staff | WIC Clients
Number analyzed (Participants) | 0 | 383
Participants
  No barriers |  | 314
  Lack of time |  | 33
  Lack of transportation |  | 32
  Unanswered |  | 4

3. Primary Outcome: Lack of Time at WIC Appointments as a Barrier to Implementing Weight Management Interventions as Described by WIC Staff
Description: WIC staff were asked to choose the how they feel about lack of time as a barrier to implementing weight management interventions at WIC appointments.
Time Frame: 1 day
Population: This question was only asked as part of the WIC staff survey as it dealt directly with barriers that WIC Staff experience.
Measure: Count of Participants; unit: Participants
Arm/Group | WIC Staff | WIC Clients
Number analyzed (Participants) | 164 | 0
Participants
  Strongly Disagree | 5 |
  Disagree | 4 |
  Neither Disagree or Agree | 19 |
  Agree | 71 |
  Strongly Agree | 61 |
  Unanswered | 4 |

4. Primary Outcome: Lack of Staff at WIC Appointments as a Barrier to Implementing Weight Management Interventions as Described by WIC Staff
Description: WIC staff were asked to choose the how they feel about lack of staff as a barrier to implementing weight management interventions at WIC appointments.
Time Frame: 1 day
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | WIC Staff | WIC Clients
Number analyzed (Participants) | 164 | 0
Participants
  Strongly Disagree | 8 |
  Disagree | 13 |
  Neither Disagree or Agree | 33 |
  Agree | 58 |
  Strongly Agree | 47 |
  Unanswered | 5 |

5. Primary Outcome: Lack of Training at WIC Appointments as a Barrier to Implementing Weight Management Interventions as Described by WIC Staff
Description: WIC staff were asked to choose the how they feel about lack of training as a barrier to implementing weight management interventions at WIC appointments.
Time Frame: 1 day
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | WIC Staff | WIC Clients
Number analyzed (Participants) | 164 | 0
Participants
  Strongly Disagree | 12 |
  Disagree | 11 |
  Neither Disagree or Agree | 23 |
  Agree | 76 |
  Strongly Agree | 37 |
  Unanswered | 5 |

ADVERSE EVENTS:
Description: Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | WIC Staff | WIC Clients
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Completeness checks were not used.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No